CLINICAL TRIAL: NCT01401790
Title: Use of a Telehomecare Program for Young Patients With New Onset Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Huot, Celine, M.D. (Other)
Responsible Party: Celine Huot MD, Centre Hospitalier Universitaire Sainte-Justine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CHUSTEJUSTINE2644
Record Dates: First submitted 2011-07-08; First posted 2011-07-25 (Estimated); Last update posted 2011-07-25 (Estimated); Status verified 2011-07

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Children; Adolescents; Telehomecare
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Telehomecare (Experimental): 3 month use of a new telehomecare program
  Interventions: Device: Telehomecare (Intelligent Distance Patient Monitoring)
- Control (Active Comparator): 3 month regular education program and follow up at the Diabetes Clinic
  Interventions: Other: Standard education and follow up at diabetes clinic

INTERVENTIONS:
Device: Telehomecare (Intelligent Distance Patient Monitoring) — Randomized patients were to be taugth and to use for 3 months a telehomecare program designed for
  * Automatic download of blood glucose levels
  * Automatic alerts indicating hypoglycemias, hyperglycemias and ketones to the medical team
  * Changes in treatment plan by the diabetes professionals
  * E mail exchanges between families and health care professionals
  * Reinforcement of teaching program
  Other Names: Telehealth; Telemonitoring
  Arms: Telehomecare
Other: Standard education and follow up at diabetes clinic — Patients allocated to the control branch receive standard diabetes teaching and care.
  Other Names: Standard diabetes care
  Arms: Control

SUMMARY:
In a Pediatric University Teaching Hospital in Montreal, an Intelligent Distance Patient Monitoring Program was developed to allow for:

* Automatic download of blood glucose levels
* Automatic alerts indicating hypoglycemias, hyperglycemias and ketones to the medical team
* Changes in treatment plan by the diabetes professionals
* E mail exchanges between families and health care professionals
* Reinforcement of teaching program

Use of this program does not replace the existing diabetes education program nor does it preclude contacts with the diabetes team. This service was devised to complement the care already in place for families of children and adolescents with diabetes, hence the term ''telehomecare-enhanced'' approach.

Hypotheses

* This approach would not incur more health problems for Web e Phone users when compared to patients treated by the ''conventional'' approach (telephone and FAX).
* Use of the Web e Phone would save time for members of the diabetes health providers and consequently cut costs.
* This means of communication would be acceptable and user friendly for both families and health care professionals.

OBJECTIVE - To determine the effects of a telehomecare (THC) program used for 3 months in families of children and adolescents with newly diagnosed type 1 diabetes.

RESEARCH DESIGN AND METHODS - A bilingual telehomecare program was developed for type 1 diabetes at the Centre Hospitalier Universitaire Sainte-Justine in Montreal. Between February 2008 and August 2009, newly diagnosed patients and their family were randomly assigned to the standard education program or to the telehomecare-enhanced group. Outcomes of interest were patients' and parents' health (reported number for total and nocturnal hypoglycemias; quality of life using the Diabetes Quality of life for Youth questionnaire and a validated Life Habits survey); knowledge of diabetes (using pre and post intervention questionnaires); organizational impacts (number and time for contacts with the nurses or with the physician on call) and family satisfaction with the software application.

DETAILED DESCRIPTION:
STUDY PROTOCOL

This is a randomized controlled study, unblinded.

The recruitment occured on Day 3 of teaching: random assignment (1:1) to receive either traditional follow up (telephone contacts and FAX communications) with the designated nurse OR a follow up with telehomecare PLUS the follow up by a specialized nurse.

If the patient is designated to telehomecare, the training is provided on day of recruitment and patient leaves with the Web e Phone. Activation of the device must be done at home to enable for transmission of information.

Families complete questionnaires to evaluate knowledge, Quality of Life Questionnaires (Skinner modified), a validated Life Habits survey and a satisfaction questionnaire at recruitment (time 0) and at study completion (3 months) (Children must be aged more than 8 years).

All reported hypoglycemias (less than 3 mmol/L) and nocturnal hypoglycemias by any means (telephone, FAX or Web e Phone) during the follow up period (suggested for 3 months) are to be accounted for.

ELIGIBILITY:
Inclusion Criteria:

* Child or adolescent with newly diagnosed type 1 diabetes

Exclusion Criteria:

* Inability to write or communicate in writing in French or English Blindness Exclusive follow up in another health center once teaching is complete

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 86 (Actual)
Dates: Start 2008-02; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Patients' health (reported number of hypoglycemias and nocturnal hypoglycemias) | 3 months
  All reported hypoglycemias (less than 3 mmol/L) by any means (telephone, FAX or Web e Phone) during the follow up period (3 months) to be accounted for in intervention and control groups

SECONDARY OUTCOMES:
Patients and parents' health | 3 months
  Families complete questionnaires to evaluate Quality of Life Questionnaires (Skinner modified) and a validated Life Habits Questionnaire at recruitment and at study completion (Children must be more than 8 years).
Knowledge of diabetes | 3 months
  using in house validated pre and post intervention questionnaires
Organizational impacts | 3 months
  Number and time required for contacts with the nurse at the clinic and / or with the physician on call
Family satisfaction with the software application | 3 months
  Using an in house validated questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec, Canada

REFERENCES:
- [Background] Chase HP, Pearson JA, Wightman C, Roberts MD, Oderberg AD, Garg SK. Modem transmission of glucose values reduces the costs and need for clinic visits. Diabetes Care. 2003 May;26(5):1475-9. doi: 10.2337/diacare.26.5.1475. PMID 12716807
- [Background] d'Annunzio G, Bellazzi R, Larizza C, Montani S, Pennati C, Castelnovi C, Stefanelli M, Rondini G, Lorini R. Telemedicine in the management of young patients with type 1 diabetes mellitus: a follow-up study. Acta Biomed. 2003;74 Suppl 1:49-55. PMID 12817805
- [Background] Izquierdo R, Morin PC, Bratt K, Moreau Z, Meyer S, Ploutz-Snyder R, Wade M, Weinstock RS. School-centered telemedicine for children with type 1 diabetes mellitus. J Pediatr. 2009 Sep;155(3):374-9. doi: 10.1016/j.jpeds.2009.03.014. Epub 2009 May 21. PMID 19464030
- [Background] Pare G, Jaana M, Sicotte C. Systematic review of home telemonitoring for chronic diseases: the evidence base. J Am Med Inform Assoc. 2007 May-Jun;14(3):269-77. doi: 10.1197/jamia.M2270. Epub 2007 Feb 28. PMID 17329725
- [Background] Rami B, Popow C, Horn W, Waldhoer T, Schober E. Telemedical support to improve glycemic control in adolescents with type 1 diabetes mellitus. Eur J Pediatr. 2006 Oct;165(10):701-5. doi: 10.1007/s00431-006-0156-6. Epub 2006 May 3. PMID 16670859
- [Background] Skinner TC, Hoey H, McGee HM, Skovlund SE; Hvidore Study Group on Childhood Diabetes. A short form of the Diabetes Quality of Life for Youth questionnaire: exploratory and confirmatory analysis in a sample of 2,077 young people with type 1 diabetes mellitus. Diabetologia. 2006 Apr;49(4):621-8. doi: 10.1007/s00125-005-0124-0. Epub 2006 Jan 26. PMID 16525844
- See also: Description of technological evaluation ongoing in institution where the project is done — http://www.chu-sainte-justine.org/Pro/Page.aspx?ID_PAGE=10002900